CLINICAL TRIAL: NCT03968939
Title: Postoperative Sleep Quality Following Total Joint Arthroplasty: A Prospective, Randomized, Controlled Trial of Diphenhydramine and Melatonin Versus Sleep Skills Training
Brief Title: Total Joint Arthroplasty and Sleep
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: James A. Keeney (Other)
Responsible Party: Sponsor-Investigator, James A. Keeney, Chief Adult Hip and Knee Reconstruction Service, Department of Orthopaedic Surgery, University of Missouri, University of Missouri-Columbia
Organization: University of Missouri-Columbia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013726
Record Dates: First submitted 2019-05-23; First posted 2019-05-30 (Actual); Results first posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-06

CONDITIONS: Primary Total Hip Arthroplasty; Primary Total Knee Arthroplasty
MeSH Terms: interventions — Diphenhydramine; Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: 1. Benadryl + Melatonin Group + Sleep Hygiene Education
  2. Sleep Hygiene Education Group
  3. Control group (Usual Care)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (Usual Care) (No Intervention): Control Group (Usual Care): Participants do not use any type of sleep education or non-prescription sleep medications to assist with getting a "good night's sleep".
- Sleep Hygiene Education (Active Comparator): Sleep Hygiene Education: Participants are provided a Sleep Hygiene Education Brochure containing information about getting a "good night's sleep."
  Interventions: Behavioral: Sleep Hygiene Education
- Over-the-counter sleep aids (25 mg Benadryl + 3mg melatonin) (Active Comparator): Participants are given both:
  1. Over-the-counter sleep aids:25 mg Diphenhydramine (Benadryl) and 3mg oral melatonin to be taken before bedtime;
  2. and a Sleep Hygiene Education Brochure containing information about getting a "good night's sleep."
  Interventions: Drug: Diphenhydramine (Benadryl); Dietary Supplement: Melatonin; Behavioral: Sleep Hygiene Education

INTERVENTIONS:
Drug: Diphenhydramine (Benadryl) — Oral Diphenhydramine (Benadryl), 25 mg
  Arms: Over-the-counter sleep aids (25 mg Benadryl + 3mg melatonin)
Dietary Supplement: Melatonin — Oral Melatonin, 3 mg
  Arms: Over-the-counter sleep aids (25 mg Benadryl + 3mg melatonin)
Behavioral: Sleep Hygiene Education — Brochure containing information about getting a "good night's sleep."
  Arms: Over-the-counter sleep aids (25 mg Benadryl + 3mg melatonin); Sleep Hygiene Education

SUMMARY:
To compare non-prescription sleep aids (low-dose diphenhydramine and melatonin) to sleep hygiene education for improving postoperative sleep quality after total joint arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

All patients undergoing elective primary total hip or knee arthroplasty

Exclusion Criteria:

1. History of substance abuse
2. Workman's compensation patients
3. Revision joint replacement
4. History of prescription or over-the- counter sleep aid use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-05-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vicki L Jones, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group (Usual Care) | Sleep Hygiene Education | Over-the-counter Sleep Aids (25 mg Benadryl + 3mg Melatonin)
Started | 15 | 26 | 14
Completed | 15 | 26 | 14
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group (Usual Care) | Sleep Hygiene Education | Over-the-counter Sleep Aids (25 mg Benadryl + 3mg Melatonin) | Total
Number analyzed (Participants) | 15 | 26 | 14 | 55
Age, Continuous [Mean (Full Range); unit: Years] | 67.77 [55 to 81] | 67.19 [53 to 80] | 66.47 [57 to 75] | 66.71 [55 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 18 | 3 | 27
  Male | 9 | 8 | 11 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 14 | 26 | 14 | 54
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 15 | 26 | 14 | 55
Total Joint Arthroplasty (TJA) Cohort [Count of Participants; unit: Participants]
  Total Knee Arthroplasty (TKA) | 9 | 18 | 9 | 36
  Total Hip Arthroplasty (THA) | 6 | 8 | 5 | 19

OUTCOME MEASURES:

1. Primary Outcome: Epworth Sleepiness Scale (ESS)
Description: Epworth Sleepiness Scale is widely used in the field of sleep medicine as a subjective measure of a patient's sleepiness. The test is a list of eight situations in which to rate the participants tendency to become sleepy.
  * No chance of dozing = 0
  * Slight chance of dozing = 1
  * Moderate chance of dozing = 2
  * High chance of dozing = 3
  Total the values of the responses. The total score is based on a scale of 0 to 24. The higher score the higher the chance the participant is experiencing excessive sleepiness.
Time Frame: Baseline, 2 weeks, 6 weeks and 12 weeks post-op
Population: Due to attrition, the number analyzed at each time point is the number of participants who followed up with the research team
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group (Usual Care) | Sleep Hygiene Education | Over-the-counter Sleep Aids (25 mg Benadryl + 3mg Melatonin)
Number analyzed (Participants) | 15 | 26 | 14
score on a scale
  Baseline | 7.73 (4.06) | 7.81 (5.04) | 8.36 (5.51)
  2 Week Follow Up: number analyzed (Participants) | 13 | 18 | 10
  2 Week Follow Up | 7.31 (3.66) | 8.17 (3.76) | 7.30 (4.67)
  6 Week Follow Up: number analyzed (Participants) | 13 | 22 | 12
  6 Week Follow Up | 8.00 (4.26) | 8.36 (4.82) | 6.17 (2.21)
  12 Week Follow Up: number analyzed (Participants) | 10 | 19 | 8
  12 Week Follow Up | 6.40 (3.17) | 6.68 (3.74) | 8.13 (6.10)

2. Primary Outcome: Pittsburgh Sleep Quality Index (PSQI)
Description: The PSQI measures several different aspects of sleep, offering seven component scores and one composite score. The component scores consist of subjective sleep quality, sleep latency (i.e., how long it takes to fall asleep), sleep duration, habitual sleep efficiency (i.e., the percentage of time in bed that one is asleep), sleep disturbances, use of sleeping medication, and daytime dysfunction.
  Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the nine component scores, providing an overall score ranging from 0 to 27, where lower scores denote a healthier sleep quality.
Time Frame: Baseline, 2 weeks, 6 weeks and 12 weeks post-op
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group (Usual Care) | Sleep Hygiene Education | Over-the-counter Sleep Aids (25 mg Benadryl + 3mg Melatonin)
Number analyzed (Participants) | 15 | 26 | 14
score on a scale
  Baseline | 10.13 (4.44) | 10.96 (4.77) | 12.14 (6.00)
  2 Weeks Follow Up: number analyzed (Participants) | 13 | 18 | 10
  2 Weeks Follow Up | 9.46 (3.97) | 13.17 (3.50) | 12.55 (5.87)
  6 Weeks Follow Up: number analyzed (Participants) | 13 | 22 | 12
  6 Weeks Follow Up | 10.38 (5.98) | 11.77 (3.46) | 6.81 (3.74)
  12 Weeks Follow Up: number analyzed (Participants) | 10 | 19 | 8
  12 Weeks Follow Up | 9.4 (3.53) | 10.7 (4.41) | 7.33 (3.64)

3. Primary Outcome: Visual Analogue Scale (VAS) for Pain
Description: Patient Reported Outcome Measure - pain Scale: 0-10. 0 being no pain and 10 being unbearable pain
Time Frame: Baseline, 2 weeks, 6 weeks and 12 weeks post-op
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group (Usual Care) | Sleep Hygiene Education | Over-the-counter Sleep Aids (25 mg Benadryl + 3mg Melatonin)
Number analyzed (Participants) | 15 | 26 | 14
score on a scale
  Baseline | 4.67 (3.04) | 4.46 (2.08) | 6.21 (1.93)
  2 Week Follow Up: number analyzed (Participants) | 13 | 18 | 10
  2 Week Follow Up | 4.31 (2.46) | 3.67 (2.00) | 4.09 (1.87)
  6 Week Follow Up: number analyzed (Participants) | 13 | 22 | 12
  6 Week Follow Up | 2.67 (1.67) | 2.36 (1.56) | 2.45 (1.81)
  12 Week Follow Up: number analyzed (Participants) | 10 | 19 | 8
  12 Week Follow Up | 1.8 (1.32) | 2.55 (1.50) | 2.78 (2.95)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent to the 12 week follow-ip
Description: The study used the definition of an adverse event defined by clinicaltrials.gov. Participants were reviewed for any untoward medical occurrences during their study participation. No adverse events were identified over the course of the study
Groups:
- Over-the-counter Sleep Aids (25 mg Benadryl + 3mg Melatonin): Participants are given both:
  1. Over-the-counter sleep aids:25 mg Diphenhydramine (Benadryl) and 3mg oral melatonin to be taken before bedtime;
  2. and a Sleep Hygiene Education Brochure containing information about getting a "good night's sleep."
  Diphenhydramine (Benadryl): Oral Diphenhydramine (Benadryl), 25 mg
  Melatonin: Oral Melatonin, 3 mg
  Sleep Hygiene Education: Brochure containing information about getting a "good night's sleep."
Arm/Group | Control Group (Usual Care) | Sleep Hygiene Education | Over-the-counter Sleep Aids (25 mg Benadryl + 3mg Melatonin)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/26 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/26 | 0/14
Other Adverse Events (participants affected / at risk) | 0/15 | 0/26 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2020-03-06): https://cdn.clinicaltrials.gov/large-docs/39/NCT03968939/Prot_000.pdf